CLINICAL TRIAL: NCT00448721
Title: A Phase II Trial of Perifosine Following Tyrosine Kinase Inhibitor Failure in Patients With Advanced Renal Cell Carcinoma
Brief Title: A Phase II Trial of Perifosine Following Tyrosine Kinase Inhibitor (TKI) - Failure in Patients With Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 228
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2012-02

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; tyrosine kinase inhibitor failure
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perifosine (Experimental): Perifosine will be administered orally at 100mg PO daily with food. One treatment cycle will consist of 42 days (6 weeks).
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — Perifosine will be administered orally at 100mg PO daily with food.
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a single-arm phase II trial of perifosine in renal cancer patients who have experienced disease progression after receiving either sorafenib or sunitinib.

DETAILED DESCRIPTION:
This is a single-arm phase II trial assessing the antitumor activity as measured by progression free survival of perifosine in patients with metastatic RCC who have progressed on sorafenib or sunitinib. A total of 48 patients will be enrolled in the trial. All subjects will have histologically confirmed metastatic RCC with predominantly clear cell features (≤ 50% other histologic features). Patients who have been taken off sorafenib or sunitinib may only have been off therapy for less than three months prior to study enrollment. Patients who remain on sorafenib or sunitinib may continue on drug at their current dose until two weeks prior to the initiation of perifosine therapy.

The study consists of three periods: pre-treatment/screening, treatment, and follow-up. Day 1 will be defined as the first day of perifosine therapy. Patients will remain in the treatment phase until progression or toxicity. Patients will be seen by an MD every 3 weeks with 6 weeks defining one cycle of therapy. Tumor evaluations will occur every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be required to have clear cell renal cell carcinoma with less than 50% of any other histology (papillary or chromophobe or oncocytic). There must be histologic confirmation by the treating center of either the primary or a metastatic lesion
* Patients must have experienced disease progression by RECIST criteria while on sorafenib or sunitinib
* Patients must be off of sorafenib or sunitinib for >= 2 weeks prior to initiation of perifosine and <= 3 months prior to enrollment
* Patients may have had sorafenib or sunitinib in the adjuvant setting as long as they have experienced disease recurrence while on therapy
* Patients must have measurable disease that is not curable by standard radiation therapy or surgery
* Age >= 18 years
* ECOG performance status 0 or 1
* - Patients must have the ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History or clinical evidence of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastasis, or history of stroke
* Other than sorafenib or sunitinib, patients may have only had prior immunotherapy for stage IV disease
* Patients may have had prior sorafenib OR sunitinib and cannot have been treated with both TKIs
* Patients who have stopped sorafenib or sunitinib due to toxicity but have only progressed off therapy will not be allowed
* Patients may have had prior anti-angiogenic such as bevacizumab only if given in combination with either sorafenib or sunitinib
* Prior Thalidomide or IFNα are allowed for adjuvant therapy or stage IV disease
* Patients may not have had prior mTOR inhibitors (CCI-779, RAD001)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To estimate the progression free survival | Every 6 weeks
  To estimate the progression free survival of Multi-Targeted Kinase Inhibitor (TKI) resistant patients with metastatic Renal Cell Carcinoma (RCC) who are treated with perifosine

SECONDARY OUTCOMES:
To determine the objective response rate of perifosine | Every 6 weeks
  To determine the objective response rate of TKI resistant patients with metastatic RCC treated with perifosine.
To investigate the tolerability and toxicity | Every 6 weeks
  To investigate the tolerability and toxicity of perifosine in TKI resistant patients
To investigate surrogates of biologic target inhibition | Every 6 weeks
  To investigate surrogates of biologic target inhibition on PBMC's before and after therapy.
To collect pre-treatment tissue specimens | Every 6 weeks
  To collect pre-treatment tissue specimens and assess the pre-treatment activation status of the MAP-Kinase and PI3K-Akt pathways and correlate with clinical outcome.
To follow levels of pro-angiogenic cytokines | Every 6 weeks
  To follow levels of pro-angiogenic cytokines and surrogates of HIF activation before and during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Investigative Site, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Nashville, Tennessee

REFERENCES:
- [Result] Journal of Clinical Oncology, 2009 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 27, No 15S (May 20 Supplement), 2009: 5101